CLINICAL TRIAL: NCT04396340
Title: A Phase 1b, First-in-Human, Dose Escalation and Expansion Study of XMT-1592 In Patients With Solid Tumors Likely to Express NaPi2b
Brief Title: First-in-Human Study of XMT-1592 in Patients With Ovarian Cancer and NSCLC Likely to Express NaPi2b
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: discontinued development program
Sponsor: Mersana Therapeutics (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMT-1592-1
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Open-label, dose escalation to reach MTD. The MTD will be confirmed in 2 parallel cohorts: (1) patients with platinum-resistant ovarian cancer; (2) patients with non-squamous NSCLC, adenocarcinoma subtype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): XMT-1592 is administered in groups of patients who will receive doses that increase over time until the maximum tolerated dose is achieved.
  Interventions: Biological: XMT-1592
- Confirmation of Dose (Experimental): New groups of patients will receive XMT-1592 at the maximum tolerated dose to confirm the recommended Phase 2 dose
  Interventions: Biological: XMT-1592

INTERVENTIONS:
Biological: XMT-1592 — XMT-1592 will be administered once every 21 or 28 days until disease progression, unacceptable toxicity, or either the patient or study physician determines it is in the best interest of the patient to discontinue participation in the study.

SUMMARY:
Phase 1b, a study in high grade serous ovarian cancer and nonsmall cell lung cancer to evaluate the safety and clinical activity of the antibody-drug conjugate (ADC) XMT-1592.

DETAILED DESCRIPTION:
This Phase 1b trial is an open-label, multi-center study of XMT-1592 administered as an intravenous infusion once every 3 weeks. The dose-escalation (DES) segment of the study will establish the expansion (EXP) dose and is intended to establish the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) for XMT-1592 in patients with high grade serous ovarian cancer (HGSOC) or non-small cell lung cancer (NSCLC), adenocarcinoma subtype. The EXP segment of the study will consist of 2 parallel cohorts of patients (HGSOC and NSCLC) to confirm the MTD or RP2D and estimate the objective response rate in each selected patient population. In DES, the observation period for dose-limiting toxicities is 21 days, between Day 1 through the end of Cycle 1 which includes the pre-dose assessments before receiving the Cycle 2 dose. All adverse events (AEs) will be graded according to NCI, CTCAE v5.0). In general, AEs ≥Grade 3 are dose-limiting toxicities with some modifications.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* ECOG performance status 0 or 1.
* Measurable disease as per RECIST, version 1.1. Resolution of all acute toxic effects of prior therapy or surgical procedures to Grade ≤1 (except alopecia).
* Adequate organ function.
* Confirmed availability of tumor tissue blocks or freshly cut tissue slides for NaPi2b testing. -In EXP, ability to undergo a fresh biopsy before enrollment, unless not medically feasible.
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective form of hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner, and to continue the use of contraception for the duration of study treatment and for at least 6 months after the last dose of study treatment.
* Histologically or cytologically confirmed solid tumors of the types specified below, with incurable, locally advanced or metastatic disease that has failed standard therapy or for which no standard treatment option exists.
* Ovarian Cancer: Histological diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal cancer, excluding the mucinous subtype.

NSCLC: Histological diagnosis of nonsquamous NSCLC.

Exclusion Criteria:

* Major surgery within 28 days of starting study treatment; -or- systemic anti-cancer therapy within the lesser of 28 days or 5 half-lives of the prior therapy before starting study treatment -or- recent radiation therapy with unresolved toxicity.
* Brain metastases that are: untreated, progressive, have required any type of major treatment, e.g., whole-brain radiation treatment, adjuvant chemotherapy, gamma knife, to control symptoms from brain metastases within 30 days of the first study treatment. Or any history of leptomeningeal metastasis.
* Current known active infection with HIV, hepatitis B virus, or hepatitis C virus.
* No prior history of liver disease such as liver cirrhosis, hepatic fibrosis
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease) or intercurrent illness that could interfere with per-protocol evaluations.
* Severe dyspnea at rest due to complications of advanced malignancy, or requiring supplementary oxygen therapy.
* Currently active pneumonitis or interstitial lung disease.
* Pregnant or nursing women.
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or other malignancy with a similar expected curative outcome.
* Participation in the DES component of the study.
* Prior use of mirvetuximab soravtansine or another ADC containing an auristatin or maytansinoid payload.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose or recommended Phase 2 dose | Up to 36 weeks, from the date of first dose until unacceptable side effects or a dose-limiting toxicity is me
  Evaluate adverse events and use of concomitant medication use after XMT-1592 doses

SECONDARY OUTCOMES:
Time of maximum observed concentration of XMT-1592 | Daily for one week after first dose; weekly until 21 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1592
Maximum concentration of XMT-1592 | Daily for one week after first dose; weekly until 21 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1592
Area under the concentration curve of the last measurable concentration of XMT-1592 | Daily for one week after first dose; weekly until 21 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1592
Antineoplastic effects of XMT-1592 | Every 6 weeks for up to 36 weeks
  Monitor tumor size
Anti-drug antibody and neutralizing antibody | Every 3 weeks for 9 weeks then every 6 weeks for upto 36 weeks
  Analyze blood for antibodies to XMT-1536 and neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burger, MD, Study Director — Mersana Therapeutics
Locations (1):
- Mary Crowley Cancer Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No